CLINICAL TRIAL: NCT02968121
Title: A Phase 1, Two-part, Open-label, Randomized, Exploratory and Single Ascending Dose, Parallel Arm Trial to Determine the Pharmacokinetics, Safety, and Tolerability of Brexpiprazole Long-acting Injectable Administered Subcutaneously or Intramuscularly in Adult Subjects With Schizophrenia
Brief Title: Safety and Tolerability Study of Single-dose Administration of Brexpiprazole in Adult Subjects With Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part A of study was completed per protocol. Conduct of Part B of the study (confirmatory phase) was not necessary.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 331-201-00033
Record Dates: First submitted 2016-11-02; First posted 2016-11-18 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: Single Dose Injection: Subcutaneous (Experimental): Drug: Brexpiprazole, OPDC-34712 Once, subcutaneous
  Interventions: Drug: Brexpiprazole, OPDC-34712
- Part A: Single Dose Injection: Intramuscular (Experimental): Drug: Brexpiprazole, OPDC-34712 Once, subcutaneous
  Interventions: Drug: Brexpiprazole, OPDC-34712
- Part B: Cohort 1 (Experimental): Drug: Brexpiprazole, OPDC-34712 Once, SC or IM
  Interventions: Drug: Brexpiprazole, OPDC-34712
- Part B: Cohort 2 (Experimental): Drug: Brexpiprazole, OPDC-34712 Once, SC or IM
  Interventions: Drug: Brexpiprazole, OPDC-34712
- Part B: Cohort 3 (Experimental): Drug: Brexpiprazole, OPDC-34712 Once, SC or IM
  Interventions: Drug: Brexpiprazole, OPDC-34712

INTERVENTIONS:
Drug: Brexpiprazole, OPDC-34712

SUMMARY:
To determine the pharmacokinetics, safety and tolerability of brexpiprazole administered subcutaneously or intramuscularly in adults with schizophrenia.

DETAILED DESCRIPTION:
This trial is designed to assess the pharmacokinetics, safety and tolerability of brexpiprazole in the treatment of subjects with schizophrenia. The trial will consist of two parts across 13-36 months. The trial population will include approximately 110 male & female subjects between 18 and 64 years of age (inclusive) with a diagnosis of schizophrenia as defined by DSM-V criteria.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 64 years of age, inclusive, at the screening visit with a diagnosis of schizophrenia as defined by DSM-V criteria.
* Body mass index between 18 and 35 kg/m^2 at the screening visit.
* Good physical health as determined by no clinically significant deviation from normal.
* Ability to provide informed consent and/or consent obtained from a legally acceptable representative (as required by IRB), prior to the initiation of any protocol-required procedures.
* Male and female subjects who are surgically sterile, female subjects who have been postmenopausal for at least 12 consecutive months prior to the screening visit, or male subjects/female subjects (of childbearing potential) who agree to remain abstinent or to practice 2 of the approved birth control methods from the screening visit and for at least 150 days after the dose of IMP for a female subject or 180 days after the dose of IMP for a male subject.

Exclusion Criteria:

* Subjects who have:
* Met DSM-V criteria for substance use disorder within the past 180 days; including alcohol and benzodiazepines, excluding caffeine/nicotine.
* A positive drug screen for drugs of abuse (excluding stimulants, other prescribed medications, and marijuana [if in investigator's documented opinion the subject does not meet DSM-V criteria for substance use disorder]).
* Use of more than 1 psychotropic medication at the screening or baseline visit, except for oral brexpiprazole administered during the brexpiprazole tolerability testing (if applicable) and current oral antipsychotic medication.
* Use of varenicline beyond screening.
* Subjects who have participated in any clinical trial involving a psychotropic medication within 1 month prior to the administration of IMP or 5 half-lives from last IMP administration whichever is longer.
* Subjects who have a significant risk of committing suicide based on history, routine psychiatric status examination, investigator's judgment, or who have an answer of "yes" on questions 4 or 5 on the Baseline Version of the C-SSRS.
* Subjects currently in an acute relapse of schizophrenia as assessed by the investigator.
* Subjects with a current DSM-V diagnosis other than schizophrenia. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Suicidality via Columbia-Suicide Severity Rating Scale | Part A: Screening to Day 182; Part B: Screening to Day 126
  Baseline version and Since Last Visit version of CSSRS will be completed by trained trial center staff
Number of reported Adverse Events (AE) | Part A: 182 days; Part B: 126 days
Clinical Laboratory Tests | Part A: 182 days; Part B: 126 days
  Hematology, serum chemistry, urinalysis, drug screen, etc. will be performed.
Change in physical exam results | Part A: Screening to Day 182; Part B: Screening to Day 126
  Investigator or designee will perform complete physical exam and document any clinically significant conditions. Body height and weight will also be measured for BMI calculation and weight will be measured as part of all subsequent physical exams.
Change in Systolic/Diastolic blood pressure from screening to end of study | Part A: Screening to Day 182; Part B: Screening to Day 126
  Heart rate and body temperature will also be obtained prior to PK blood draws and ECG.
ECG Reading | Part A: 182 days; Part B: 126 days
  12-lead ECG will be collected in triplicate (5 minutes apart). heart rate, ventricular rate, RR interval, PR interval, QRS duration and QT intervals will be recorded. QTcF and corrected QT interval using Bazett's formula will be calculated.
Extrapyramidal Symptoms (EPS) Rating Scale | Part A: 182 days; Part B: 126 days
  SAS, AIMS & BARS will be assess by trained trial center staff
Investigator's assessment of injection site | Part A: 182 days; Part B: 126 days
  Injection site will be assessed. Injection site will also be inspected for seepage after needle is withdrawn.
Visual analog scale (VAS) scores for pain reception | Part A: 182 days; Part B: 126 days

SECONDARY OUTCOMES:
Maximum peak plasma concentration (Cmax) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411.
Time of Cmax (tmax) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411
Area under the concentration-time curve (AUC) from time zero to time "t" (Last observable concentration; AUCt) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411
AUC from time zero to infinity (AUC∞) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411
Terminal-phase elimination half-life (t1/2,z) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411
Apparent clearance of drug from plasma after extravascular administration (CL/F; brexpiprazole only) [Pharmacokinetics] | Day 1 (predose [within 2 hours prior to dosing] and 4, 8 , and 12 hours postdose)
  Samples will also be collected on Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112, 126, 154, and 182/ET or until plasma concentrations of brexpiprazole are BLQ, whichever is longer based on monthly PK sampling (samples will be collected between 8 AM and 2 PM on the indicated nondosing day). If a PK blood sample cannot be drawn at the designated time on Day 1, a window of ± 15 minutes for each blood draw is acceptable with the exact time recorded.
  PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) including DM-3411

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuro Science (CNS), Garden Grove, California
  - CNRI, San Diego, California